CLINICAL TRIAL: NCT04674488
Title: An Exploratory Clinical Study of TILs Treatment for Metastatic or Recurrent Cervical Cancer
Brief Title: TILs for Treatment of Metastatic or Recurrent Cervical Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai OriginCell Therapeutics Co., Ltd. (Industry)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OriginCell
Record Dates: First submitted 2020-12-13; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: TILs, Metastatic or Recurrent Cervical Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TILs intervention (Experimental)
  Interventions: Biological: TILs

INTERVENTIONS:
Biological: TILs — a single center, single-arm, open label, interventional study

SUMMARY:
Prospective, single center, single-arm, open label, interventional study evaluating adoptive cell therapy (ACT) with autologous tumor infiltrating lymphocytes (TIL) infusion followed by IL-2 after a non-myeloablative (NMA) lymphodepletion preparative regimen for the treatment of patients with recurrent, metastatic cervical carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years old;
2. ECOG (Eastern Cooperative Oncology Group) score is 0 or 1;
3. The case is diagnosed as cervical squamous cell carcinoma, adenosquamous carcinoma or cervical adenocarcinoma;
4. Patients who have metastasized or relapsed after initial treatment (surgery, chemotherapy or radiotherapy);
5. HPV (Human Papillomavirus)-DNA test shows HPV16 positive and/or HPV18 positive;
6. At least one measurable target lesion defined by RECIST v1.1 (Response Evaluation Criteria in Solid Tumours);
7. The subject must have a lesion with a diameter of more than 10 mm and a volume of 1.5 cm3 or more (or a collection of resected lesions greater than or equal to 1.5 cm3). TILs can be separated after resection or malignant effusion;
8. Routine blood testing reaches the following indicators: neutrophils ≥ 1.5×10^9/L, PLT ≥60×10^9/L, Hb ≥9.0 g/dL, LY ≥0.4×10^9/L;
9. Liver and kidney function: ALT (Alanine Aminotransferase, alanine aminotransferase) or AST (Aspartate Aminotransferase, aspartate aminotransferase) index <2.5 times the normal value; creatinine clearance rate>50 ml/min; total bilirubin <1.5 times the normal value, Prothrombin time prolonged ≤ 4 s;
10. The treatment methods for malignant tumors, including radiotherapy, chemotherapy and biological agents (including granulocyte colony stimulating factor G-CSF, targeted drug therapy, etc.), must be stopped 28 days before the TILs are obtained;
11. Subjects with reproductive potential must be willing to implement the approved high-efficiency contraceptive method with informed consent and continue to implement it within 1 year after the completion of the clinical trial;
12. The subject is able to adhere to the research visit plan and other protocol requirements.

Exclusion Criteria:

1. Uncontrolled active systemic infection; patients with active viral hepatitis;
2. Confirmed HIV infection;
3. The electrocardiogram indicates myocardial ischemia; the left ventricular ejection fraction on ultrasonography of subjects over 40 years old is less than 45%;
4. Pulmonary function test (spirometry) proves that forced expiratory volume (FEV) 1<65% predicted or forced vital capacity (FVC)<65% predicted;
5. Patients with a history of COPD (Chronic Obstructive Pulmonary Disease), asthma, or other chronic lung diseases with significant symptoms;
6. The subject received systemic steroids equivalent to >15 mg/day of prednisone 2 weeks before sampling, except for inhaled steroids;
7. The patient has hereditary or acquired coagulopathy;
8. Medical history of organ or hematopoietic stem cell transplantation;
9. Patients who are pregnant or breastfeeding;
10. Those who suffer from serious neurological, mental or endocrine diseases, or those who have serious mental diseases that will hinder full informed consent;
11. The medical history of primary immunodeficiency, past immune system diseases includes autoimmune diseases that are active, or previously known or suspected to exist autoimmune diseases. Except for side effects of checkpoint inhibitors, vitiligo, psoriasis, type 1 diabetes, remission of childhood asthma, and remission of atopic side effects.
12. Suffered from other uncured malignant tumors in the past 5 years or at the same time, except skin basal cell carcinoma and thyroid cancer.
13. There are central nervous system metastases and central nervous system diseases with clinical significance;
14. Live vaccine was vaccinated 30 days before cell reinfusion;
15. Patients with a previous history of cell therapy within one year;
16. Patients with a history of acute drug allergy, especially those who are allergic to immunoglobulin drugs;
17. Any other conditions judged by the researcher will significantly increase the risk of participation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-11-09 (Estimated); Study Completion 2024-11-09 (Estimated)

PRIMARY OUTCOMES:
dose limited toxicity, DLT | 28 days
  Safety and tolerability of TILs, as determined by the rate of Dose Limiting Toxicities (DLTs)

SECONDARY OUTCOMES:
Objective Response Rate, ORR | three months
  To evaluate the efficacy of TILs in patients with recurrent, metastatic cervical carcinoma based on the objective response rate (ORR) as assessed by the Independent Review Committee (IRC) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Duration of Response, DOR | two years
  To evaluate the efficacy parameters of TILs in patients with recurrent, metastatic cervical carcinoma by assessing duration of response (DOR) as assessed by the IRC per RECIST v1.1
Progression-Free Survival, PFS | two years
  To evaluate the efficacy parameters of TILs in patients with recurrent, metastatic cervical carcinoma by assessing progression-free survival (PFS) as assessed by the IRC per RECIST v1.1
overall survival, OS | two years
  To evaluate overall survival (OS) in patients with recurrent, metastatic cervical carcinoma
Disease Control Rate, DCR | two years
  To evaluate the efficacy of TILs in patients with recurrent, metastatic cervical carcinoma by assessing disease control rate (DCR) as assessed by the Investigator per RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai general hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
to publish papers